CLINICAL TRIAL: NCT05759364
Title: The Effect of IV PAPAVERINE 80 mg Prior to Catheter Balloon Insertion on Bishop Score and Pain, Double Blinded Randomized Placebo Controlled Trial
Brief Title: The Effect of IV PAPAVERINE 80 mg Prior to Catheter Balloon Insertion on Bishop Score and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Director of Maternal-fetal medicine, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0012-23-NHR
Record Dates: First submitted 2023-02-14; First posted 2023-03-08 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Induction of Labor; Pain, Acute; Labor Pain; Delivery Delayed
Keywords: Induction of labor; Ripenning of the cervix; Catheter balloon; Antispasmodic
MeSH Terms: conditions — Acute Pain; Labor Pain | interventions — Papaverine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blinded randomized placebo controlled trial Group 1: will get IV PAPAVERINE 80 mg in 100 ml saline Group 2: will get IV 100 ml saline
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant will be blinded to the type of therapy they recieved. Inverstiagators will be blinded. Outcome assessor, including the physican that will assess the bishop score will be blinded Only the nurse that gives the therapy won't be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- IV PAPAVERINE 80 mg (Active Comparator): Administration of IV PAPAVERINE 80 mg in 100 ml of saline, once within half an hour before inserting a single-balloon balloon catheter
  Interventions: Drug: IV Papaverine 80 mg
- Conrol group- Placebo group. (Placebo Comparator): Administration of 100 ml of saline within half an hour before the insertion of a single-balloon catheter
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Papaverine 80 mg — Opium alkaloid antispasmodic drug
  Other Names: Papaverine Hydrochloride
  Arms: Intervention group- IV PAPAVERINE 80 mg
Drug: Placebo — Placebo
  Other Names: Saline
  Arms: Conrol group- Placebo group.

SUMMARY:
The cervix consists of connective tissue, smooth muscle, and parasympathetic innervation. Smooth muscle makes up about 15% of the cervix, is mainly found under the internal opening of the neck. Papaverine and its derivatives are musculotropic antispasmodic drugs that directly affect smooth muscle, the mechanism is to reduce the spasm of smooth muscle resulting in relaxation. Studies on the pharmacokinetics of this drug show that it has a half-life of 0.5-2 hours and its effect is apparent within 10 minutes.

Administration of antispasmodic drugs during childbirth is common in developing and developed countries. Based on previous studies, the use of these drugs during childbirth may lead to a faster opening of the cervix. Possible uses of Papaverine include, administered separately or in combination with other treatments such as rupture of amniotic membranes and/or Oxytocin administration. According to some studies, administration of Papaverine at birth can be used as a preventive or therapeutic strategy in cases of prolonged labor or first stage over 12 hours as defined in some studies. According to Kochran et al, who included 13 experiments with 1995 participants, the use of antispasmodic drugs shortened the first stage of labor by an average of 74.34 minutes. In 6 experiments that included 820 patients, the administration of antispasmodic drugs during labor increases the rate of cervical opening by an average of 0.61 cm per hour.

In addition to the muscle relaxation effect, studies have been published on the analgesic effect of PAPAVERINE for example in patients with urinary stones.

In the present study, the investigators want to test the effect of administering PAPAVERINE IV 80 mg within half an hour before the insertion of a catheter balloon for cervical ripening on the Bishop score after catheter removal between the two groups.

DETAILED DESCRIPTION:
There are different methods of induction of labor, the choice of the best method for that patient depends on the bishop score, an estimate that is based on data related to the cervix such as opening, effacement and other parameters, also the choice of the method of induction depends on the obstetric history of the patient. A Bishop score less than 6 indicates an unriped cervix, therefore increasing the chance of labor induction failure,methods have been developed to ripen the cervix; among the methods are catheter balloon insertion and prostaglandins. The mechanisms by which the catheter works include a mechanical effect and indirect effect on local secretion of prostaglandins.

The cervix consists of connective tissue, smooth muscle, and parasympathetic innervation. Smooth muscle makes up about 15% of the cervix, is mainly found under the internal opening of the neck. Papaverine and its derivatives are musculotropic antispasmodic drugs that directly affect smooth muscle, the mechanism is to reduce the spasm of smooth muscle resulting in relaxation. Studies on the pharmacokinetics of this drug show that it has a half-life of 0.5-2 hours and its effect is apparent within 10 minutes.

Administration of antispasmodic drugs during childbirth is common in developing and developed countries. Based on previous studies, the use of these drugs during childbirth may lead to a faster opening of the cervix. Possible uses of Papaverine include, administered separately or in combination with other treatments such as rupture of amniotic membranes and/or Oxytocin administration. According to some studies, administration of Papaverine at birth can be used as a preventive or therapeutic strategy in cases of prolonged labor or first stage over 12 hours as defined in some studies. According to Kochran et al, who included 13 experiments with 1995 participants, the use of antispasmodic drugs shortened the first stage of labor by an average of 74.34 minutes. In 6 experiments that included 820 patients, the administration of antispasmodic drugs during labor increases the rate of cervical opening by an average of 0.61 cm per hour.

In addition to the muscle relaxation effect, studies have been published on the analgesic effect of PAPAVERINE for example in patients with urinary stones.

In the present study, the investigators want to test the effect of administering PAPAVERINE IV 80 mg within half an hour before the insertion of a catheter balloon for cervical ripening on the Bishop score after catheter removal between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton pregnancy, over the age of 18, pregnant at term (ie between weeks 37-42)
* Bishop score is less than 6, for which a medical decision was made regarding the induction of labor by catheter
* Vertex presentation, intact membranes
* Viable fetus

Exclusion Criteria:

* Twin pregnancy
* Women after caesarean section
* Severe fetal anomalies
* Women with vaginismus or vulvodynia
* Women with psychiatric illnesses including depression and schizophrenia
* Contraindication for vaginal delivery
* A woman who is unable to sign a consent form
* Women are known for supraventricular tachycardia
* Women with tachycardia over 100 or arrhythmia
* Known sensitivity to one of the components of the drug
* Liver disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Obstetrical research
Enrollment: 128 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The delta Bishop score | 1 year
  The difference between the bishop score (a score of the cervix ripening) before and after the insertion of Foley catheter. Higher delta Bishop scores means better outcome
Pain during insertion of the catheter | 1 year
  Pain during insertion of the catheter based on visual scale analoug (0-10) score, . The minimum is 0, the maximum is 10. Higher score means worse outcome

SECONDARY OUTCOMES:
Induction-delivery interval | 2 years
  Time from insertion of the catheter balloon to delivery. Longer interval means worse outcome
Success | 2 years
  Bishop score (a score of cervix ripenining) after extraction of the catheter above or equal to 8. Bishop score above or equal to 8, means better outcome
Use of other ripening method | 2 years
  The need for other ripening method due to low bishop score (<6) after extraction of the catheter balloon
Insertion-extraction of the catheter interval | 2 years
  Time between insertion to extraction of the catheter balloon.
Delivery method | 2 years
  Cesarean or vaginal delivery
Maternal satisfaction | 1 year
  Based on visual scale analoug score for satisfaction (1-5), the minimum is 1, the maximum is 5, higher score means better outcome
Apgar Score | 2 years
  The Apgar score, is a score given to the newborn in 1,5 and 10 minutes after birth, and is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth.
Cord pH | 2 years
  Cord blood gas analysis is an objective measure of the fetal metabolic condition at the time of delivery
Need for neonatal intensive case admission | 2 years
  Is a measure of neonatal complications at birth

CONTACTS AND LOCATIONS:
Overall Officials: Maya Frank Wolf, MD, Principal Investigator — Galilee Medical Center
Locations (1):
- Galilee Medical Center, Nahariya, Northern District, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rohwer AC, Khondowe O, Young T. Antispasmodics for labour. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD009243. doi: 10.1002/14651858.CD009243.pub2. PMID 22895986
- [Background] Singh KC, Jain P, Goel N, Saxena A. Drotaverine hydrochloride for augmentation of labor. Int J Gynaecol Obstet. 2004 Jan;84(1):17-22. doi: 10.1016/s0020-7292(03)00276-5. PMID 14698825
- [Background] Ibrahim MI, Alzeeniny HA, Ellaithy MI, Salama AH, Abdellatif MA. Drotaverine to improve progression of labor among nulliparous women. Int J Gynaecol Obstet. 2014 Feb;124(2):112-7. doi: 10.1016/j.ijgo.2013.08.013. Epub 2013 Nov 7. PMID 24299975
- [Background] Madhu C, Mahavarkar S, Bhave S. A randomised controlled study comparing Drotaverine hydrochloride and Valethamate bromide in the augmentation of labour. Arch Gynecol Obstet. 2010 Jul;282(1):11-5. doi: 10.1007/s00404-009-1188-8. Epub 2009 Jul 31. PMID 19644697
- [Background] Snir N, Moskovitz B, Nativ O, Margel D, Sandovski U, Sulkes J, Livne PM, Lifshitz DA. Papaverine hydrochloride for the treatment of renal colic: an old drug revisited. A prospective, randomized study. J Urol. 2008 Apr;179(4):1411-4. doi: 10.1016/j.juro.2007.11.053. Epub 2008 Mar 4. PMID 18289563
- [Derived] Abu Shqara R, Nakhleh Francis Y, Goldinfeld G, Haddad Y, Sgayer I, Lavinsky M, Lowenstein L, Frank Wolf M. Papaverine prior to catheter balloon insertion for labor induction: a randomized controlled trial. Am J Obstet Gynecol MFM. 2024 Jul;6(7):101388. doi: 10.1016/j.ajogmf.2024.101388. Epub 2024 May 31. PMID 38825005